CLINICAL TRIAL: NCT07281196
Title: A Real-World Study on Changes in Sleep Apnea Among Patients With Type 2 Diabetes/Obesity and Comorbid OSA After Short-Term Treatment With Semaglutide
Brief Title: Semaglutide Effects on Sleep Apnea in Patients With Type 2 Diabetes/Obesity and Comorbid Obstructive Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Shanghai Fengxian District Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-KY-56-02
Record Dates: First submitted 2025-11-19; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-08

CONDITIONS: Sleep Apnea Syndrome (OSAS)
Keywords: Semaglutide; Type 2 Diabetes; GLP-1 receptor agonist; real-world study; metabolic syndrome; AHI
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Semaglutide Treatment Group: single-arm cohort of 15 patients with T2DM/obesity and OSA receiving semaglutide(0.25-2.4mg/week) for 4 weeks
  Interventions: Drug: Semaglutide Subcutaneous Injection

INTERVENTIONS:
Drug: Semaglutide Subcutaneous Injection — This study is a observational study and the treatments are based on the clinical practice. In the study, patients with treatments were recorded. According to the instructions of drugs, 1ml of the injection contains 1.34mg of semaglutide. Each pre-filled injection pen contains 2mg of semaglutide and is placed in 1.5ml of solution. This product should be injected once a week.

SUMMARY:
Semaglutide (a GLP-1RA) is approved for type 2 diabetes mellitus T2DM and obesity, but its effect on obstructive sleep apnea OSA remains unclear.

To evaluate changes in Apnea-Hypopnea Index (AHI) after 1-week and 4-week semaglutide treatment in T2DM/obesity patients with OSA, we conducted a single-center real-world study (RWS) of 15 patients. Outcomes assessed included AHI, weight, BMI, blood pressure, blood glucose(fasting blood glucose, glycated albumin),liver function, blood lipids, waist circumference, and other metabolic parameters, to provide real-world evidence for semaglutide in OSA management.

DETAILED DESCRIPTION:
1. Background Obesity (BMI ≥27 kg/m²) affects over 2.2 billion adults globally and exacerbates comorbidities including cardiovascular disease(CVD), obstructive sleep apnea (OSA) and type 2 diabetes mellitus (T2DM). Semaglutide, a GLP-1 receptor agonist(GLP-1RA), demonstrates significant weight loss (5-20% at 2.4 mg/week) and metabolic benefits in trials. Emerging evidence suggests it may improve OSA by reducing central respiratory dysregulation. However, real-world data on its short-term effects on AHI remain scarce.
2. Objectives Primary: Assess change in apnea-hypopnea index (AHI) after 1-week semaglutide treatment.

   Secondary:

   AHI change at 4 weeks. Weight, BMI, waist circumference, blood pressure, glucose (fasting glucose, glycated albumin), liver function, and lipids at 1 and 4 weeks.
3. Study Design Type: Single-center observational real-world study. Data Source: Structured electronic medical records (EMR) from Fengxian Central Hospital.
4. Study Population 4.1 Inclusion Criteria:

(1) Age 18-65 years. (2) BMI ≥27 kg/m²,with ≥1 comorbidity (hypertension, dyslipidemia, CVD) or T2DM.

(3) On the basis of dietary control and exercise, the therapeutic effect is not satisfactory. There are indications for the use of semaglutide in clinical practice.

(4) Combined with obstructive sleep apnea syndrome. (5) Within the past month, no hormone drug treatment that affects glucose and lipid metabolism, nor any drugs such as antibiotics that significantly interfere with the oral flora, or bariatric surgery has been received。 (6) With complete information for this study. 4.2 Exclusion Criteria.

1. Abnormal weight gain caused by endocrine diseases (pituitary/adrenal diseases, such as Cushing's syndrome; Or hypothyroidism, etc.)
2. Severe renal/hepatic impairment (eGFR <45 mL/min; ALT/AST >2.5×ULN).
3. Severe metabolic diseases, such as diabetic ketoacidosis and hyperosmolar hyperglycemic state, etc.
4. Patients with type 1 diabetes or other special types of diabetes, patients with type 2 diabetes with severely impaired pancreatic islet function, or patients with type 2 diabetes who use insulin.
5. There is a known history of drug use that affects glycolipid metabolism within three months, such as ① glucocorticoids; ② Fluoroquinolone antibiotics; ③ Beta-blockers such as metoprolol, etc. ④ Thyroid preparations such as thyroid hormone tablets; ⑤ Psychotropic drugs, including antipsychotic drugs such as chlorpromazine and olanzapine, as well as anti-anxiety or anti-depression drugs like SSRIS and NaSSAs; ⑥ SABA bronchodilators such as salbutamol and terbutaline; ⑦ Other known drugs that affect glycolipid metabolism, such as statins.
6. Severe bleeding tendency, urinary and reproductive system infections; There are contraindications for the use of semaglutide, such as a history of acute or chronic pancreatitis, medullary thyroid carcinoma, and multiple endocrine neoplasia (MEN) type 2.
7. Patients with contraindications to radiological examinations.
8. Patients with advanced malignant tumors.
9. Severe cardiovascular and cerebrovascular diseases, such as heart failure, etc.
10. Rheumatic immune diseases, etc.
11. Pregnant women and lactating women.
12. Patients who have taken or are currently taking diuretics such as loop diuretics and thiazides within the past month.
13. Currently involved in other interventional researchers.
14. Other situations that the researchers consider unsuitable for the study, such as poor compliance, etc.

5. Treatment Records 5.1 Drug: Semaglutide subcutaneous injection. 5.2 Dosing: 1ml of the injection contains 1.34mg of semaglutide. Each pre-filled injection pen contains 2mg of semaglutide and is placed in 1.5ml of solution. This product should be injected once a week. It can be administered at any time of the day without the need to follow meal times. This product is administered by subcutaneous injection. The injection site can be selected from the abdomen, thigh or upper arm. There is no need to adjust the dosage when changing the injection site. In all cases, patients should resume a regular weekly dosing schedule.

5.3 Concomitant Medications: The patient's medical records should detail the situation of concomitant medication during the study period and must comply with the management regulations for the concomitant medication of semaglutide In particular, metformin, sulfonylurea drugs, glucocorticoids, fluoroquinolone antibiotics, beta-blockers such as metoprolol, thyroid preparations such as thyroid hormone tablets, psychotropic drugs, anti-anxiety or anti-depression drugs such as SSRIS and NaSSAs, SABA bronchodilators, and other known drugs that affect glucose and lipid metabolism should be recorded.

6. Endpoints

The study will evaluate the following endpoints:

6.1 Primary Endpoint: Change in AHI measured by PSG from baseline (T0) to 1 week post-treatment (T1).

6.2 Secondary Endpoints:

1. Changes in weight (units: kg), from T0 to T1 and 2 weeks post-treatment (T2);
2. Changes in BMI, from T0 to T1 and T2;
3. waist circumference (units: cm), from T0 to T1 and T2;
4. blood pressure (units: mmHg), from T0 to T1 and T2;
5. Changes in metabolic markers from T0 to T1 and T2 inlcuding

   * fasting glucose (mmol/L)

     * glycated albumin (%) ③ liver enzymes (U/L)

       * lipid profiles (mmol/L)

         7. Statistical Analyses 7.1 Sample Size Estimation 15 patients (80% power, α=0.05, paired Wilcoxon Signed-Rank test; anticipated ΔAHI=-10.58±10 from pilot data).

7.2 Data Handling Missing Data: Patients with missing baseline or follow-up AHI measurements will be excluded from the primary analysis.

Outliers: Values outside the 95% normal range will be reviewed for potential data entry errors or biological plausibility before analysis.

7.3 Primary Analyses The primary endpoint (sleep PSG parameters) was compared with the baseline treatment at 4 weeks after treatment using the paired rank sum test to assess whether the change was statistically significant. If the P value was less than 0.05, it could be considered that the sleep PSG parameters had decreased after treatment. Other secondary endpoint indicators (liver function, blood glucose, etc.) were also compared with baseline treatment at 4 weeks after treatment using the paired rank sum test to assess whether the change was statistically significant. If the P value was less than 0.05, it could also be considered that there was a change.

7.4 Secondary Analyses If the dosage of medication for some patients is adjusted during the study period, subgroup analyses will be conducted based on different doses. For instance, if the first dose is 0.25mg and then adjusted to 0.5mg or maintained at 0.25mg, further analysis will be conducted in different subgroups.

7.5 Sensitivity Analyses To assess the stability of the research results, external controls, published data, and data from other patients treated concurrently will be introduced for evaluation, and the differences before and after treatment will be compared. To minimize the impact of outliers, data outside the 95% range will be presented during the analysis to assess the consistency of the results. For some doses that are inconsistent, the results will be evaluated through inclusion and exclusion, and the consistency will be compared.

7.6 Quality control The quality control of this study consists of two parts. The data collected in the retrospective study must ensure the completeness of the data and the consistency of the equipment. The data collected in the prospective study will be subject to quality control on the standardization of the CRF table, the parameters of the equipment, and the operators to avoid measurement errors caused by human or equipment factors.

8. Ethics Approved by Fengxian Central Hospital (IRB No.：2025-KY-56-02) De-identified EMR data extracted under broad consent for secondary research. Compliance with China's Personal Information Protection Law (PIPL).

9. Timeline Data collection: Jan 2025-Dec 2025. Analysis: Jan 2026. Study completion: 31-Jan-2026.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years. 2. BMI ≥27 kg/m²,with ≥1 comorbidity (hypertension, dyslipidemia, CVD) or T2DM. 3. On the basis of dietary control and exercise, the therapeutic effect is not satisfactory. There are indications for the use of semaglutide in clinical practice.

4. Combined with obstructive sleep apnea syndrome. 5. Within the past month, no hormone drug treatment that affects glucose and lipid metabolism, nor any drugs such as antibiotics that significantly interfere with the oral flora, or bariatric surgery has been received.

6. With complete information for this study. Exclusion Criteria.

1. Abnormal weight gain caused by endocrine diseases (pituitary/adrenal diseases, such as Cushing's syndrome; Or hypothyroidism, etc.)
2. Severe renal/hepatic impairment (eGFR <45 mL/min; ALT/AST >2.5×ULN).
3. Severe metabolic diseases, such as diabetic ketoacidosis and hyperosmolar hyperglycemic state, etc.
4. Patients with type 1 diabetes or other special types of diabetes, patients with type 2 diabetes with severely impaired pancreatic islet function, or patients with type 2 diabetes who use insulin.
5. There is a known history of drug use that affects glycolipid metabolism within three months, such as ① glucocorticoids; ② Fluoroquinolone antibiotics; ③ Beta-blockers such as metoprolol, etc. ④ Thyroid preparations such as thyroid hormone tablets; ⑤ Psychotropic drugs, including antipsychotic drugs such as chlorpromazine and olanzapine, as well as anti-anxiety or anti-depression drugs like SSRIS and NaSSAs; ⑥ SABA bronchodilators such as salbutamol and terbutaline; ⑦ Other known drugs that affect glycolipid metabolism, such as statins.
6. Severe bleeding tendency, urinary and reproductive system infections; There are contraindications for the use of semaglutide, such as a history of acute or chronic pancreatitis, medullary thyroid carcinoma, and multiple endocrine neoplasia (MEN) type 2.
7. Patients with contraindications to radiological examinations.
8. Patients with advanced malignant tumors.
9. Severe cardiovascular and cerebrovascular diseases, such as heart failure, etc.
10. Rheumatic immune diseases, etc.
11. Pregnant women and lactating women.
12. Patients who have taken or are currently taking diuretics such as loop diuretics and thiazides within the past month.
13. Currently involved in other interventional researchers.
14. Other situations that the researchers consider unsuitable for the study, such as poor compliance, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 adults with T2DM/obesity and OSA receiving semaglutide
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Apnea-Hypopea Index(AHI) | Baseline and 1 week
  Absolute change in AHI from baseline to 1 week after semaglutide treatment

SECONDARY OUTCOMES:
Changes in weight | Baseline, 1 week, 4 weeks
  Absolute change in body weight (kg) from baseline to 1 and 4 weeks.
Changes in BMI | Baseline, 1 week, 4 weeks
  Absolute change in BMI (kg/m2) from baseline to 1 and 4 weeks.
Changes in waist circumference | Baseline, 1 week, 4 weeks
  Absolute change in waist circumference (cm) from baseline to 1 and 4 weeks.
Changes in blood pressure | Baseline, 1 week, 4 weeks
  Absolute change in blood pressure (mmHg) from baseline to 1 and 4 weeks.

OTHER OUTCOMES:
Changes in fasting glucose | baseline,1 week,4 weeks
  absolute changes in fasting glucose (mmol/L), from baseline to T1 and T2.
Changes in glycated albumin | baseline,1 week,4 weeks
  absolute changes in glycated albumin (%), from baseline to T1 and T2.
Changes in liver enzymes | baseline,1 week,4 weeks
  absolute changes in liver enzymes (U/L), from baseline to T1 and T2.
Changes in lipid profiles | baseline,1 week,4 weeks
  absolute changes in lipid profiles (mmol/L), including total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol from baseline to T1 and T2.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Fengxian District Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: World Obesity Atlas 2024 | World Obesity Federation[EB/OL]. [2024-10-28] — https://www.worldobesity.org/